CLINICAL TRIAL: NCT07222956
Title: An Open-label, Single-center Study of Remibrutinib Using Ultra High-field (7T) MR Imaging in Relapsing or Progressive MS (RemiSeven)
Brief Title: A Study of Remibrutinib Using MR Imaging in Relapsing or Progressive MS
Acronym: RemiSeven
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Moein Amin (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Moein Amin, Principal Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RS-001
Record Dates: First submitted 2025-10-23; First posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Multiple Sclerosis (MS) - Relapsing-remitting; Multiple Sclerosis (MS) Secondary Progressive; Multiple Sclerosis (MS) Primary Progressive
Keywords: multiple sclerosis; Relapsing; Progressive; Remibrutinib
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis; Recurrence | interventions — remibrutinib

STUDY DESIGN:
Intervention Model Description: investigator-run, open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Remibrutinib, active administration (Experimental): 100 mg remibrutinib, twice daily
  Interventions: Drug: Remibrutinib (Open Label)

INTERVENTIONS:
Drug: Remibrutinib (Open Label) — 100 mg remibrutinib, twice daily

SUMMARY:
The study is an investigator-run, study following participants for 2 years with twice-daily remibrutinib. MRI is the main endpoint. Safety, tolerability, and efficacy are secondary endpoints. Approximately 20 participants with relapsing or progressive forms of MS will be recruited.

DETAILED DESCRIPTION:
The study is an investigator-run, open-label Phase 2 study with approximately 24 total months of observation, involving approximately 20 participants with relapsing or progressive forms of MS.

Participants will be recruited from the patient populations followed at CCF. All participants will take 100 mg remibrutinib twice daily. They will receive 4 MRIs, blood tests, EKGs, physical exams, and clinical functioning exams periodically to assess safety, tolerability, and efficacy of the study drug. All study activities will be performed at the Cleveland Clinic Mellen Center.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, participants must meet the following eligibility criteria at the Screening visit:

1. Written informed consent signed by participant.
2. English-speaking.
3. Male and female participants, 18-60 years of age inclusive.
4. Established diagnosis of relapsing or progressive MS, as defined by the 2024 revision of McDonald Diagnostic Criteria (any form of MS). A diagnosis of MS must be confirmed at the time of the screening visit.
5. Expanded Disability Status Score (EDSS) of 0 - 6.5, inclusive.
6. Adequate vision and motor function to participate in assessment procedures.
7. Females participating in the study must meet one the following criteria:

   1. Surgically sterilized (e.g., hysterectomy, bilateral oophorectomy or tubal ligation) for at least 6 months or postmenopausal (postmenopausal females must have no menstrual bleeding for at least 1 year) or
   2. If not postmenopausal, agree to use a double method of contraception, one of which is a barrier method (e.g., intrauterine device plus condom, spermicidal gel plus condom) 30 days prior to dosing until 30 days after last dose and have negative human chorionic gonadotropin (β-hCG) test for pregnancy at screening and at each follow-up visit.
8. Males who have not had a vasectomy must use appropriate contraception methods (barrier or abstinence) from 30 days prior to dosing until 30 days after last dose.
9. Evidence of disease activity in the prior 12 months (at least one clinical relapse or one gadolinium enhancing lesion or new T2 lesion) or presence of disability worsening based clinician's assessment in the prior 12 months.
10. Participants should be in reasonably good health and neurologically stable over the last 1 month (no MS relapse in this period).

Exclusion Criteria:

Participants will be excluded from the study if any of the following exclusion criteria exist at the Screening Visit:

1. Concurrent treatment with any disease modifying therapy for MS or systemic immunotherapy for other autoimmune or rheumatological disorders (e.g. rheumatoid arthritis, systemic lupus erythematosus, inflammatory bowel disease) according to study protocol.
2. Ongoing substance abuse (drug or alcohol) or any other factor that may interfere with the participant's ability to cooperate and comply with study procedures.
3. History of malignancy of any organ system (other than complete resection of localized basal cell carcinoma of the skin or in situ cervical cancer) within the past 5 years regardless of treatment or metastasis status.
4. History of liver disease or liver function abnormalities at baseline including Gilbert syndrome.
5. History of severe renal disease or creatinine level above 1.5 x upper limit normal.
6. Pregnancy, planned or current.
7. History of severe depression or suicidality.
8. Hematological abnormalities at screening: hemoglobin < 10 g/dl, platelets < 100000/mm3, absolute lymphocyte count < 800/mm3, white blood cells < 3000/mm3, neutrophils < 1500/mm3, B-cell count < 50% lower limit of normal, total IgG or total IgM < lower limit of normal.
9. Active clinically significant bacterial, viral, parasitic, or fungal infections, in the judgement of the investigator.
10. History of significant central nervous system disease (e.g. stroke, traumatic brain injury, myelopathy, progressive multifocal leukoencepahalopathy).
11. History of splenectomy.
12. History of active or latent tuberculosis with a positive QuantiFERON, at screening.
13. Individuals with a known immunodeficiency syndrome, drug-induced immunodeficiency, hereditary immunodeficiency, or who test positive for Human immunodeficiency virus (HIV) antibody, at screening
14. Clinically significant cardiovascular, renal, hepatic, endocrine, metabolic, hematological, pulmonary, or gastrointestinal disorders that in the investigator's opinion would compromise the safety of the participant or interfere with the interpretation of the study results.
15. History or current diagnosis of ECG abnormalities such as concomitant clinically significant cardiac arrhythmias, history of familial long QT syndrome, cardiac arrhythmias requiring anti-arrhythmic treatment with class Ia or III anti-arrhythmic drugs.
16. Resting QT interval corrected by Fridericia's formula (QTcF) >450 msec (male) or >460 msec (female) prior to screening.
17. Requirement for anticoagulant medication or use of dual anti-platelet therapy. Use of acetylsalicylic acid up to 100 mg/day or clopidogrel up to 75 mg/day, is permitted.
18. Significant bleeding risk or history of clinically significant bleeding disorders.
19. Use of gastric acid modifying agents, such as proton pump inhibitors or H2 antagonists.
20. Use of any strong inhibitors of CYP3A4 (including clarithromycin, grapefruit, itraconazole, ketoconazole), or strong or moderate inducers of CYP3A4 (including carbamazepine, phenytoin, St John's Wort, primidone, modafinil). Concomitant medicines will be examined on a case-by-case basis.
21. Live vaccines within 6 weeks prior to screening or requirement to receive these vaccinations at any time during study treatment.
22. Inability to complete MRI with contrast (claustrophobia, pacemaker, cochlear implant, metallic implants incompatible with MR, hypersensitivity to gadolinium-based contrast agent, or severe renal disease).
23. Other factors that the Investigator determines would place the individual at risk for participation or interfere with interpretation of the results.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-10-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Quantitative MRI volumetric measurements | Baseline to Month 24
  Rate of change in regional brain volumes using 7T MRI over 24 months
Slowly expanding lesions (SELs) | Baseline to Month 24
  Prevalence of SELs identified using 7T MRI over 24 months
Paramagnetic rim lesions (PRLs) -- count | Baseline to Month 24
  Change in count of PRLs identified using 7T MRI over 24 months
Paramagnetic rim lesions (PRLs) -- size | Baseline to Month 24
  Change in size of PRLs identified using 7T MRI over 24 months
Paramagnetic rim lesions (PRLs) -- quantitative susceptibility measures | Baseline to Month 24
  Change in quantitative susceptibility measures of PRLs identified using 7T MRI over 24 months
Myelin Water Fraction | Baseline to Month 24
  Rate of change in myelin water fraction assessed using 7T MRI over 24 months
Functional MRI (Default mode network) | Baseline to Month 24
  Functional MRI changes (default mode network) assessed using 7T MRI over 24 months
Microstructural tissue integrity | Baseline to Month 24
  Rate of change in microstructural tissue integrity assessed using 7T MRI over 24 months
Leptomeningeal enhancement | Baseline to Month 24
  Prevalence of leptomeningeal enhancement identified using 7T MRI over 24 months
Neuromelanin | Baseline to Month 24
  Prevalence of regional neuromelanin changes identified using 7T MRI over 24 months

SECONDARY OUTCOMES:
Frequency of Treatment Emergent Adverse Events (TEAEs) | Baseline to Month 24
Frequency of Serious Adverse Events (SAEs) | Baseline to Month 24
Frequency of study medication discontinuation | Baseline to Month 24
Gadolinium Enhancing Lesions | Baseline to Month 24
  Change in number of Gadolinium enhancing lesions over 24 months
Quantitative Lesion Burden | Baseline to Month 24
  Change in the volume of brain lesions identified over 24 months
Annualized Relapse Rate (ARR) | Baseline to Month 24
Expanded Disability Status Scale (EDSS) | Baseline to Month 24
  A scale from 0 to 10. An increase in EDSS score is indicative of an increase in disability
Serum Neurofilament Light Chain (NfL) | Baseline to Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Moein Amin, MD, MS, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided